CLINICAL TRIAL: NCT03373058
Title: A Phase III Multicenter Prospective Randomized Controlled Clinical Trial of Hyperthermic Intraperitoneal Chemotherapy in the Treatment of Advanced-Stage Epithelial Ovarian Cancer After Cytoreductive Surgery
Brief Title: Efficacy of HIPEC in the Treatment of Advanced-Stage Epithelial Ovarian Cancer After Cytoreductive Surgery
Acronym: EHTASEOCCS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Henan Provincial People's Hospital (Other); Xiangya Hospital of Central South University (Other); The Third Xiangya Hospital of Central South University (Other); Peking University Cancer Hospital & Institute (Other); Peking University People's Hospital (Other); Cancer Hospital of Guizhou Province (Other); Chinese PLA General Hospital (Other); Hebei Medical University Fourth Hospital (Other); The Second Hospital of Hebei Medical University (Other); West China Second University Hospital (Other); Peking Union Medical College Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Henan Cancer Hospital (Other Government); Tianjin Medical University Cancer Institute and Hospital (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other); Wuhan University (Other); RenJi Hospital (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Southern Medical University, China (Other); Fourth Affiliated Hospital of Guangxi Medical University (Other); Shandong Cancer Hospital and Institute (Other); Beijing Obstetrics and Gynecology Hospital (Other); Chongqing University Cancer Hospital (Other); Xinqiao Hospital of Chongqing (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); First Affiliated Hospital of Chongqing Medical University (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC-03
Record Dates: First submitted 2017-12-04; First posted 2017-12-14 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Hyperthermic Intraperitoneal Chemotherapy; Advanced-Stage Epithelial Ovarian Cancer; Cytoreductive surgery; Postoperative Chemotherapy
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Cytoreduction Surgical Procedures; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 1. Cytoreductive surgery
  2. Hyperthermic Intraperitoneal Chemotherapy (HIPEC) with Docetaxel 75 mg/m^2 and cisplatin 75 mg/m^2 intraperitoneally in succession
  3. 6 cycles of adjuvant chemotherapy: paclitaxel 175 mg/m^2 IV>3 hour(Docetaxel 75 mg/m^2, if paclitaxel is not available.)+ carboplatin AUC = 5-6 IV>1 hour, every 3 weeks.
  Interventions: Procedure: Hyperthermic Intraperitoneal Chemotherapy; Procedure: cytoreductive surgery; Drug: adjuvant chemotherapy
- Control group (Active Comparator): 1. Cytoreductive surgery
  2. 6 cycles of adjuvant chemotherapy: paclitaxel 175 mg/m^2 IV>3 hour(Docetaxel 75 mg/m^2, if paclitaxel is not available)+ carboplatin AUC = 5-6 IV>1 hour, every 3 weeks.
  Interventions: Procedure: cytoreductive surgery; Drug: adjuvant chemotherapy

INTERVENTIONS:
Procedure: Hyperthermic Intraperitoneal Chemotherapy — HIPEC is performed as postoperative chemotherapy after cytoreductive surgery for advanced-stage epithelial ovarian cancer. The first HIPEC is conducted within 48h after cytoreductive surgery: Paclitaxel 175 mg/m^2, 43°C, 90min. The second HIPEC is performed after 48 hours of the first HIPEC. The HIPEC regimens are Docetaxel 75 mg/m^2 and cisplatin 75 mg/m^2, respectively, 43°C, 90min.
  Other Names: HIPEC
  Arms: Experimental group
Procedure: cytoreductive surgery — Cytoreductive surgery (CRS) is performed when Faggoti value is less than 6 via laparoscopic exploration.
  Other Names: CRS
Drug: adjuvant chemotherapy — Systemic chemotherapy regimens after HIPEC treatment are paclitaxel 175 mg/m^2 IV>3 hour+ carboplatin AUC = 5-6 IV>1 hour, every 3 weeks for 2 cycles in experimental group.
  Systemic chemotherapy regimens after IDS are paclitaxel 175 mg/m^2 IV>3 hour+ carboplatin AUC = 5-6 IV>1 hour, every 3 weeks for 3 cycles in control group.
  Other Names: ACT

SUMMARY:
This project is a multi-center, prospective, randomized controlled clinical observation the safety and efficacy of hyperthermic intraperitoneal chemotherapy in the treatment of advanced-stage epithelial ovarian cancer after cytoreductive surgery. Median recurrence-free survival is the primary end points of this project.

DETAILED DESCRIPTION:
The current standard treatment for epithelial ovarian cancer, tubal cancer, and primary peritoneal cancer is maximal cytoreductive surgery followed by intravenous chemotherapy with or without intraperitoneal chemotherapy (IP). Recently, the organizations of SGO and ASCO recommended that women with Fagotti score by laparoscopic exploration < 6 would benefit from primary cytoreductive surgery followed by postoperative chemotherapy, and are likely to attain optimal cytoreduction (residual lesion ≤ 1 cm).

Hyperthermia promotes chemotherapy to penetrate deeper into the cancer tissue. Therefore, hyperthermic intraperitoneal chemotherapy (HIPEC) as newly postoperative chemotherapy after primary cytoreductive surgery in the treatment of ovarian cancer could lead to higher response rate and better survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Disease status primary epithelial ovarian cancer, tubal cancer, and primary peritoneal cancer (Stage III )
* Fagotti score by laparoscopic exploration < 6
* Residual tumor < 1cm after completion of cytoreductive surgery
* 18 < Age < 70 year old
* Expected survival > 3 months
* Performance status: ECOG 0-1
* Adequate bone marrow function Hb ≥8 g/dl (After correction in case of iron deficient anemia) WBC ≥ 3,000/mm3, Platelet ≥ 100,000/mm3
* Adequate renal function Creatinine ≤ 1.5 mg/dl, and adequate hepatic function Bilirubin ≤ 1.5 mg/dl and AST and ALT ≤ 80 IU/L
* Voluntary participation after getting written informed consent.

Exclusion Criteria:

* Fagotti score by laparoscopic exploration >= 6
* Suboptimal debulking (residual tumor > 1cm)
* Extensive adhesion in peritoneal cavity
* Previous History of other malignancies (except excision of skin cancer, thyroid cancer)
* Poorly controlled disease e.g. atrial fibrillation, stenocardia, cardiac insufficiency, persistent hypertension despite medicinal treatment, ejection fraction<50%
* Receiving other chemotherapy, radiotherapy or immunotherapy
* Patients who are unsuitable candidates by doctor's decision
* Without given written informed consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Median recurrence-free survival | 3 years
  assess median recurrence-free survival during 3 years in both study arms

SECONDARY OUTCOMES:
Median overall survival | 3 years
  assess median overall survival during 3 years in both study arms
Median progression-free survival | 3 years
  assess median progression-free survival during 3 years in both study arms
Risk factors for morbidity and mortality | 30 days; 3 years
  The early complication and mortality are defined as the event observed within 30 days after intervention, while the time frame for late complication is the period beyond 30 days after intervention to the end of 3 years. Complications are ranked from grade 0-5 according to CTCAE V4.0
Quality of life for ovarian cancer | 3 years
  Evaluated according to European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Ovarian Cancer Module (QLQ-OV28)

CONTACTS AND LOCATIONS:
Overall Officials: Shuzhong Cui, M.D, Study Director — Affiliated Cancer Hospital & Institute of Guangzhou Medical University; Zhongqiu Lin, M.D, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (7):
- China (7):
  - Affiliated Tumor Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital,Sun Yat-sen University, Guanzhou, Guangdong
  - Beijing Cancer Hospital, Beijing
  - Chongqing Cancer Hospital, Chongqing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Hubei General Hospital, Wuhan
  - Henan Cancer Hospital, Zhengzhou